CLINICAL TRIAL: NCT06589856
Title: Does Oral Lactate Affect Gut Hormone Secretion in a Dose-response Relationship?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jens Hohwü Voigt, MD, PhD student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LAMETA-DOSE-RESPONSE
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized single-blinded, placebo-controlled crossover study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CTR (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: LAC5; Dietary Supplement: LAC10; Dietary Supplement: LAC20
- LAC5 (Experimental)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: LAC5; Dietary Supplement: LAC10; Dietary Supplement: LAC20
- LAC10 (Experimental)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: LAC5; Dietary Supplement: LAC10; Dietary Supplement: LAC20
- LAC20 (Experimental)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: LAC5; Dietary Supplement: LAC10; Dietary Supplement: LAC20

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo (300 mL salt water, NaCl) = CTR
Dietary Supplement: LAC5 — 5 g lactate (300 mL lactate drink = 5 g D/L-lactate bound to Na) = LAC5
Dietary Supplement: LAC10 — 10 g lactate (300 mL lactate drink = 10 g D/L-lactate bound to Na) = LAC10
Dietary Supplement: LAC20 — 20 g lactate (300 mL lactate drink = 20 g D/L-lactate bound to Na) = LAC20

SUMMARY:
To investigate whether there is a linear dose-response relationship between oral lactate and its effects on gut hormone secretion, motility, and appetite.

Hypothesis Oral lactate administration affects gut hormone secretion, insulin levels, motility, appetite sensation and the amount of food intake in a linear dose-response relationship.

DETAILED DESCRIPTION:
The participants will meet up fasting at the Steno Diabetes Centre Aarhus Research Lab. Immediately after arrival, they will be placed in a bed. The four trial days will be completely alike, besides the interventions.

The participants will have one intravenous (iv.) access placed in the elbow on the four trial days for a continuous drawing of blood samples throughout the trial day.

Before drinking the intervention, baseline blood samples will be drawn. Immediately after drinking the intervention, the participants will take 1500 mg paracetamol to determine ventricular emptying rate through the acetaminophen test.

After this, the participants can lay in their bed and watch TV, Ipad or work on their computer. Blood samples will be collected at 0, 10, 20, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 240 minutes after the intervention. Appetite sensations will be measured by a visual analog scales (VAS). After 3 hours the trial day is finished, and the participants can go home.

Before and after each trial day the participants will collect a fecal sample.

We will use ANOVA and mixed model regression analyses for comparing the four groups.

Based on a previous study we will need 11 individuals to detect a difference of 17,3 pmol/L in mean insulin concentrations at time 60 minutes, with a SD of 18,3 (α=0.05, β=0.80). To account for potential missing values, we will include a total of 12 participants

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Written and oral consent
* Healthy

Exclusion Criteria:

* HbA1c > 39
* Taking medicine
* Any diseases
* Allergy to paracetamol
* Doesn't speak or understand Danish.
* Special diets

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean insulin concentration | 60 minutes
  Difference in mean insulin concentration 60 minutes after the intervention between CTR and LAC5, LAC10, and LAC20.

SECONDARY OUTCOMES:
Difference in blood glucose | 0-180 minutes after the intervention
Difference in GLP-1 | 0-180 minutes after the intervention
Difference in GIP | 0-180 minutes after the intervention
Difference in LEAP2 | 0-180 minutes after the intervention
Difference in glucagon | 0-180 minutes after the intervention
Difference in c-peptide | 0-180 minutes after the intervention
Difference in gastric emptying rate | 0-180 minutes after the intervention
  Acetaminophen test
Difference in appetite sensation | 0-180 minutes
  VAS (visual analoge scale)

CONTACTS AND LOCATIONS:
Overall Officials: Esben Sondergaard, Principal Investigator — Aarhus University, Steno Diabetes Center Aarhus
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided